CLINICAL TRIAL: NCT06218485
Title: Comparison of Fractional Flow Reserve-Guided Strategy Versus Intravascular Ultrasound-Guided Stent Implantation After Angiography-Derived Fractional Flow Reserve-based Decision-Making (The FLAVOUR III Trial)
Brief Title: FFR Versus IVUS with Angiography-Derived FFR for Clinical Outcomes in Patients with Coronary Artery Disease
Acronym: FLAVOUR III
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Seoul National University Hospital (Other); Peking University Third Hospital (Other); RenJi Hospital (Other); Second Affiliated Hospital of Shantou University Medical College (Other); The First Affiliated Hospital of Nanchang University (Other); First Affiliated Hospital of Kunming Medical University (Other); The Fourth People's Hospital of Jinan (Unknown); Jinhua Central Hospital (Other); The Affiliated Hospital of Hangzhou Normal University (Other); Changxing People's Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); The Affiliated Hospital of Medical College, Ningbo University (Other); Keimyung University Dongsan Medical Center (Other); Inje University Ilsan Paik Hospital (Other); Ulsan University Hospital (Other); Uijeongbu Eulji Medical Center (Unknown); Kyungpook National University Hospital (Other); Seoul St. Mary's Hospital (Other); Yonsei University Wonju Severance Hospital (Unknown); Inje University Haeundae Paik Hospital (Other); Sejong General Hospital (Other); Chonnam National University Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); The Affiliated Hospital of Shandong University of TCM (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0896
Record Dates: First submitted 2023-11-27; First posted 2024-01-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease
Keywords: Angiography-derived fractional flow reserve; Intravascular ultrasound; Fractional flow reserve; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The percutaneous coronary intervention will be performed by intravascular ultrasound (IVUS)-guided strategy after angiography-derived FFR-based decision-making.
  Interventions: Procedure: Intravascular ultrasound-guided stent implantation after angiography-derived FFR-based decision-making
- Control group (Active Comparator): The percutaneous coronary intervention will be performed by fractional flow reserve (FFR)-guided strategy.
  Interventions: Procedure: Fractional flow reserve-guided PCI strategy

INTERVENTIONS:
Procedure: Intravascular ultrasound-guided stent implantation after angiography-derived FFR-based decision-making — The percutaneous coronary intervention will be performed by intravascular ultrasound (IVUS)-guided strategy after angiography-derived FFR-based decision-making:
  1. PCI will be performed if angiography-derived FFR ≤0.80 and will be deferred if angiography-derived FFR >0.80.
  2. If PCI is performed, PCI optimization using IVUS will be performed following the recommended criteria: ① Plaque burden at stent edge ≤55%; ② Minimal stent area ≥ 5.5 mm2, or minimal stent area ≥ distal reference lumen area
  Arms: Experimental group
Procedure: Fractional flow reserve-guided PCI strategy — The percutaneous coronary intervention will be performed by fractional flow reserve (FFR)-guided strategy:
  1. PCI will be performed if FFR ≤0.80 and will be deferred if FFR >0.80.
  2. If PCI is performed, PCI optimization using FFR will be performed following the recommended criteria: ① Post-PCI FFR ≥ 0.88, or ② Post-PCI ΔFFR ([FFR at stent distal edge] - [FFR at stent proximal edge]) < 0.05
  Arms: Control group

SUMMARY:
To compare the clinical outcomes of fractional flow reserve (FFR)-guided strategy versus intravascular ultrasound (IVUS)-guided stent implantation after angiography-derived FFR-based decision-making.

DETAILED DESCRIPTION:
1. Hypothesis: The IVUS-guided stent implantation after angiography-derived FFR-based decision-making will show superiority in terms of a lower rate of patients-oriented composite outcomes (POCO) at 24 months after randomization compared with the FFR-guided PCI strategy in patients with coronary stenosis.
2. Research materials and indication for revascularization:

   2.1 Experimental group: PCI will be performed if angiography-derived FFR ≤0.80 and will be deferred if angiography-derived FFR >0.80; If PCI is performed, PCI optimization using IVUS will be performed following the recommended criteria: ① Plaque burden at stent edge ≤55%; ② Minimal stent area ≥ 5.5 mm2, or minimal stent area ≥ distal reference lumen area.

   2.2 Control group: PCI will be performed if FFR ≤0.80 and will be deferred if FFR >0.80; If PCI is performed, PCI optimization using FFR will be performed following the recommended criteria: ① Post-PCI FFR ≥ 0.88, or ② Post-PCI ΔFFR ([FFR at stent distal edge] - [FFR at stent proximal edge]) < 0.05.
3. Sample size: In the post-hoc analysis of the FLAVOUR I study applying QFR analysis, the 2-year POCO rate was 13.0% in the PCI group with FFR ≤0.80 and undergoing FFR-based PCI optimization and 7.1% in the PCI group with QFR ≤0.80 and undergoing IVUS-based PCI optimization. Meanwhile, the 2-year POCO rate was 5.8% and 6.5% in the deferral of PCI group with FFR >0.80 and QFR >0.80, respectively. Assuming a PCI rate of 70% in patients with coronary artery lesions with 50-90% stenosis that is the inclusion criteria for the current study, and considering event rates from historical studies evaluating FFR- and QFR-guided PCI strategies, the cumulative incidence rate of POCO at 24 months was estimated to be 13.0% in the control group (FFR group) and 9.0% in the experimental group (QFR-IVUS group).

   * Primary endpoint: POCO, defined as a composite of death from any cause, MI, or any revascularization at 24 months after randomization.
   * Design: superiority
   * Sampling ratio: experimental group : control group = 1:1
   * Type I error (α): One-sided 2.5%
   * Accrual time: 24 months
   * Total time: 4 years (accrual 24 months + follow-up 24 months)
   * Assumption: POCO 13.0% vs. 9.0% in control or experimental group, respectively
   * Statistical power (1- β): 90%
   * Primary statistical method: Kaplan-Meier survival analysis with log-rank test
   * Estimated attrition rate: total 10%
   * Stratification in randomization: Presence of diabetes mellitus

Based on the above assumption, we would need total 1,942 patients (971 patients in each group) with consideration of an attrition rate.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 19 years.
* Subject is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving invasive physiologic or imaging evaluation and PCI with a drug-eluting stent (DES) and he/she or his/her legally authorized representative provides written informed consent.
* Subjects suspected with ischemic heart disease.
* Subjects with coronary artery diameter stenosis 50-90% by angiography-based visual estimation eligible for stent implantation.
* Target vessel size ≥ 2.5mm in visual estimation.

Exclusion Criteria:

* Known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Prasugrel, Ticagrelor
* Active pathologic bleeding.
* Gastrointestinal or genitourinary major bleeding within the prior 3 months.
* History of bleeding diathesis, known coagulopathy.
* Non-cardiac co-morbid conditions with life expectancy < 2 years.
* Target lesion located in coronary arterial bypass graft.
* Left main coronary artery stenosis ≥ 50%.
* Chronic total occlusion in the study target vessel.
* Culprit lesion of ST-elevation myocardial infarction (STEMI).
* Not eligible for angiography-derived FFR (ostial RCA ≥ 50% stenosis, severe tortuosity, severe overlap, poor image quality).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1942 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient-oriented composite outcome | 24 months
  Patient-oriented composite outcome (POCO), defined as a composite of all death, myocardial infarction (MI), or any revascularization at 24 months after randomization.

SECONDARY OUTCOMES:
Patient-oriented composite outcome at 60 months | 60 months
  Patient-oriented composite outcome (POCO), defined as a composite of all death, myocardial infarction (MI), or any revascularization.
Individual component of Patient-oriented composite outcome | 24 and 60 months
  Individual component of Patient-oriented composite outcome (death, myocardial infarction, revascularization).
Target vessel failure | 24 and 60 months
  Target vessel failure, defined as a composite of cardiac death, target-vessel MI, or target vessel revascularization.
Cost-effectiveness analysis | 24 and 60 months
  Incremental cost effectiveness ratio (ICER).
All-cause and cardiac death | 24 and 60 months
  All-cause and cardiac death.
Any nonfatal myocardial infarction without peri-procedural myocardial infarction | 24 and 60 months
  Any nonfatal myocardial infarction without peri-procedural myocardial infarction.
Any nonfatal myocardial infarction with peri-procedural myocardial infarction | 24 and 60 months
  Any nonfatal myocardial infarction with peri-procedural myocardial infarction.
Any target vessel/lesion revascularization | 24 and 60 months
  Any target vessel/lesion revascularization.
Any non-target vessel/lesion revascularization | 24 and 60 months
  Any non-target vessel/lesion revascularization.
Any revascularization (ischemia-driven or all) | 24 and 60 months
  Any revascularization (ischemia-driven or all).
Stent thrombosis (definite/probable/possible) | 24 and 60 months
  Stent thrombosis at 24 and 60 months after randomization.
Stroke (ischemic and hemorrhagic) | 24 and 60 months
  Stroke at 24 and 60 months after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, MD, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (25):
- China (14):
  - Peking University Third Hospital, Beijing
  - Second Affiliated Hospital of Shantou University Medical College, Guangdong
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Changxing People's Hospital, Huzhou
  - The Affiliated Hospital of Shandong University of TCM, Jinan
  - The Fourth People's Hospital of Jinan, Jinan
  - Jinhua Central Hospital, Jinhua
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - The Affiliated Hospital of Medical College, Ningbo University, Ningbo
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - The First Affiliated hospital of Wenzhou Medical University, Wenzhou
- South Korea (11):
  - Bucheon Sejong Hospital, Bucheon-si
  - Inje University Haeundae Paik Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hospital, Donggu
  - Inje University Ilsan Paik Hospital, Goyang
  - Seoul National University Hospital,, Seoul
  - Seoul ST. Mary's Hospital, Seoul
  - Uijeongbu Eulji Medical Center, Uijeongbu-si
  - Ulsan University Hospital, Ulsan
  - Yonsei University Wonju Severance Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: Yes
The deidentified data will be shared after publication of first manuscript
Supporting Information: Study Protocol
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Background] Kogame N, Ono M, Kawashima H, Tomaniak M, Hara H, Leipsic J, Andreini D, Collet C, Patel MR, Tu S, Xu B, Bourantas CV, Lerman A, Piek JJ, Davies JE, Escaned J, Wijns W, Onuma Y, Serruys PW. The Impact of Coronary Physiology on Contemporary Clinical Decision Making. JACC Cardiovasc Interv. 2020 Jul 27;13(14):1617-1638. doi: 10.1016/j.jcin.2020.04.040. PMID 32703589
- [Background] Writing Committee Members; Lawton JS, Tamis-Holland JE, Bangalore S, Bates ER, Beckie TM, Bischoff JM, Bittl JA, Cohen MG, DiMaio JM, Don CW, Fremes SE, Gaudino MF, Goldberger ZD, Grant MC, Jaswal JB, Kurlansky PA, Mehran R, Metkus TS Jr, Nnacheta LC, Rao SV, Sellke FW, Sharma G, Yong CM, Zwischenberger BA. 2021 ACC/AHA/SCAI Guideline for Coronary Artery Revascularization: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2022 Jan 18;79(2):e21-e129. doi: 10.1016/j.jacc.2021.09.006. Epub 2021 Dec 9. PMID 34895950
- [Background] Raber L, Mintz GS, Koskinas KC, Johnson TW, Holm NR, Onuma Y, Radu MD, Joner M, Yu B, Jia H, Meneveau N, de la Torre Hernandez JM, Escaned J, Hill J, Prati F, Colombo A, di Mario C, Regar E, Capodanno D, Wijns W, Byrne RA, Guagliumi G; ESC Scientific Document Group. Clinical use of intracoronary imaging. Part 1: guidance and optimization of coronary interventions. An expert consensus document of the European Association of Percutaneous Cardiovascular Interventions. Eur Heart J. 2018 Sep 14;39(35):3281-3300. doi: 10.1093/eurheartj/ehy285. PMID 29790954
- [Background] De Maria GL, Garcia-Garcia HM, Scarsini R, Hideo-Kajita A, Gonzalo Lopez N, Leone AM, Sarno G, Daemen J, Shlofmitz E, Jeremias A, Tebaldi M, Bezerra HG, Tu S, Lemos PA, Ozaki Y, Dan K, Collet C, Banning AP, Barbato E, Johnson NP, Waksman R. Novel Indices of Coronary Physiology: Do We Need Alternatives to Fractional Flow Reserve? Circ Cardiovasc Interv. 2020 Apr;13(4):e008487. doi: 10.1161/CIRCINTERVENTIONS.119.008487. Epub 2020 Apr 16. PMID 32295416
- [Background] Scoccia A, Tomaniak M, Neleman T, Groenland FTW, Plantes ACZD, Daemen J. Angiography-Based Fractional Flow Reserve: State of the Art. Curr Cardiol Rep. 2022 Jun;24(6):667-678. doi: 10.1007/s11886-022-01687-4. Epub 2022 Apr 18. PMID 35435570
- [Background] Collet C, Onuma Y, Sonck J, Asano T, Vandeloo B, Kornowski R, Tu S, Westra J, Holm NR, Xu B, de Winter RJ, Tijssen JG, Miyazaki Y, Katagiri Y, Tenekecioglu E, Modolo R, Chichareon P, Cosyns B, Schoors D, Roosens B, Lochy S, Argacha JF, van Rosendael A, Bax J, Reiber JHC, Escaned J, De Bruyne B, Wijns W, Serruys PW. Diagnostic performance of angiography-derived fractional flow reserve: a systematic review and Bayesian meta-analysis. Eur Heart J. 2018 Sep 14;39(35):3314-3321. doi: 10.1093/eurheartj/ehy445. PMID 30137305
- [Background] Fearon WF, Achenbach S, Engstrom T, Assali A, Shlofmitz R, Jeremias A, Fournier S, Kirtane AJ, Kornowski R, Greenberg G, Jubeh R, Kolansky DM, McAndrew T, Dressler O, Maehara A, Matsumura M, Leon MB, De Bruyne B; FAST-FFR Study Investigators. Accuracy of Fractional Flow Reserve Derived From Coronary Angiography. Circulation. 2019 Jan 22;139(4):477-484. doi: 10.1161/CIRCULATIONAHA.118.037350. PMID 30586699
- [Background] Xu B, Tu S, Qiao S, Qu X, Chen Y, Yang J, Guo L, Sun Z, Li Z, Tian F, Fang W, Chen J, Li W, Guan C, Holm NR, Wijns W, Hu S. Diagnostic Accuracy of Angiography-Based Quantitative Flow Ratio Measurements for Online Assessment of Coronary Stenosis. J Am Coll Cardiol. 2017 Dec 26;70(25):3077-3087. doi: 10.1016/j.jacc.2017.10.035. Epub 2017 Oct 31. PMID 29101020
- [Background] Koo BK, Hu X, Kang J, Zhang J, Jiang J, Hahn JY, Nam CW, Doh JH, Lee BK, Kim W, Huang J, Jiang F, Zhou H, Chen P, Tang L, Jiang W, Chen X, He W, Ahn SG, Yoon MH, Kim U, Lee JM, Hwang D, Ki YJ, Shin ES, Kim HS, Tahk SJ, Wang J; FLAVOUR Investigators. Fractional Flow Reserve or Intravascular Ultrasonography to Guide PCI. N Engl J Med. 2022 Sep 1;387(9):779-789. doi: 10.1056/NEJMoa2201546. PMID 36053504
- [Background] Gotberg M, Christiansen EH, Gudmundsdottir IJ, Sandhall L, Danielewicz M, Jakobsen L, Olsson SE, Ohagen P, Olsson H, Omerovic E, Calais F, Lindroos P, Maeng M, Todt T, Venetsanos D, James SK, Karegren A, Nilsson M, Carlsson J, Hauer D, Jensen J, Karlsson AC, Panayi G, Erlinge D, Frobert O; iFR-SWEDEHEART Investigators. Instantaneous Wave-free Ratio versus Fractional Flow Reserve to Guide PCI. N Engl J Med. 2017 May 11;376(19):1813-1823. doi: 10.1056/NEJMoa1616540. Epub 2017 Mar 18. PMID 28317438